CLINICAL TRIAL: NCT01464437
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Explore Dose Effect and Frequency of Administration of AMG 151 in Subjects With Type 2 Diabetes Mellitus
Brief Title: AMG 151 Amgen Protocol Number 20100761
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20100761
Record Dates: First submitted 2011-10-14; First posted 2011-11-03 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; mellitus; metformin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- AMG 151 - Arm 1 (Active Comparator): AMG 151 - Arm 1
  Interventions: Drug: AMG 151; Drug: Metformin
- AMG 151 - Arm 2 (Active Comparator): AMG 151 - Arm 2
  Interventions: Drug: Metformin; Drug: AMG 151
- AMG 151 - Arm 3 (Active Comparator): AMG 151 - Arm 3
  Interventions: Drug: Metformin; Drug: AMG 151
- AMG 151 - Arm 4 (Active Comparator): AMG 151 - Arm 4
  Interventions: Drug: Metformin; Drug: AMG 151
- AMG 151 - Arm 5 (Active Comparator): AMG 151 - Arm 5
  Interventions: Drug: Metformin; Drug: AMG 151
- AMG 151 - Arm 6 (Active Comparator): AMG 151 - Arm 6
  Interventions: Drug: Metformin; Drug: AMG 151
- Placebo Arm (Placebo Comparator): AMG 151 Placebo Arm
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: AMG 151 — Drug: AMG 151 50 mg BID
  Arms: AMG 151 - Arm 1
Drug: Placebo — Placebo
  Arms: Placebo Arm
Drug: Metformin — Subjects will remain on their metformin regimen throughout the study. The metformin dose must be ≥ 850 mg/day for at least 2 months immediately prior to randomization.
Drug: AMG 151 — Drug: AMG 151 100 mg BID
  Arms: AMG 151 - Arm 2
Drug: AMG 151 — Drug: AMG 151 200 mg BID
  Arms: AMG 151 - Arm 3
Drug: AMG 151 — Drug: AMG 151 100 mg QD
  Arms: AMG 151 - Arm 4
Drug: AMG 151 — Drug: AMG 151 200 mg QD
  Arms: AMG 151 - Arm 5
Drug: AMG 151 — Drug: AMG 151 400 mg QD
  Arms: AMG 151 - Arm 6

SUMMARY:
This is a phase 2a, multicenter, randomized, double-blind, placebo-controlled, parallel group, fixed dose study. AMG 151 will be evaluated in subjects with type 2 diabetes treated with metformin for at least 3 months prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, inclusive
* Diagnosis of type 2 diabetes mellitus
* HbA1c levels 7.5% to 11.0%, inclusive, at screening
* Fasting C-peptide levels ≥ 0.2 nmol/L at screening
* BMI ≥ 25 to < 45 kg/m2 at screening
* Treated with metformin monotherapy for at least 3 months prior to randomization; the metformin dose must be ≥ 850 mg daily for at least 2 months immediately prior to randomization
* If a subject is being treated for hyperlipidemia or hypertension they should be on stable medication for 30 days before randomization
* Subject has provided informed consent.

Exclusion Criteria:

* History of type 1 diabetes
* History of significant weight gain or loss (> 10%) during the 4 weeks before randomization
* Use of any weight loss medication (over the counter or prescription) within 60 days of randomization
* Use of any oral or injectable anti-hyperglycemic medication (other than metformin) within 3 months prior to randomization
* Use of chronic and/or continuous insulin administration for > 15 days in an outpatient setting to achieve and maintain glycemic control prior to randomization
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months
* Have had more than 1 episode of severe hypoglycemia within 6 months prior to entry into the study, or currently diagnosed as having hypoglycemia unawareness
* Evidence of active infections that can interfere with the study
* Presence of clinically significant organ system disease that is not stabilized or may interfere with the study
* Currently receiving immunosuppressive therapy
* History of positive HIV, chronic hepatitis B or C, or cirrhosis
* Have symptomatic congestive heart failure or a history of myocardial infarction, unstable angina, or decompensated congestive heart failure or stroke in the past 6 months prior to screening.
* History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption
* Any finding on the screening ECG that in the opinion of the investigator requires further cardiovascular evaluation
* Poorly controlled hypertension defined as diastolic pressure > 100 mm Hg or systolic pressure > 160 mm Hg (assessed on two separate occasions during the screening period)
* Malignancy (other than resected cutaneous basal or cutaneous squamous cell carcinoma, or treated in situ cervical cancer considered cured) within 5 years of screening visit (if a malignancy occurred > 5 years ago, subject is eligible with documentation of disease-free state since treatment)
* Use of known inhibitors or inducers of CYP3A4 are not permitted 30 days prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose-effect relationship of AMG 151 compared to placebo on fasting plasma glucose in subjects with type 2 diabetes treated with metformin | Change in fasting plasma glucose levels from baseline to Day 28

SECONDARY OUTCOMES:
To assess the effect of AMG 151 on postprandial glucose levels in response to a meal tolerance test | Change in area under the curve from 0-4 hours (AUC0-4hr) glucose after a meal tolerancetest from baseline to Day 28, Change in incremental AUC0-4hr glucose after a meal tolerance test from baseline to Day 28
Adverse events | Incidence of serious adverse events from signing of ICF to Day 42. Incidence of non-serious adverse events from randomization to Day 42.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (69):
- United States (60):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Chula Vista, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Inglewood, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Desert, California
  - Research Site, Roseville, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Walnut Creek, California
  - Research Site, Watsonville, California
  - Research Site, Bradenton, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Maitland, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chigago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Metairie, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Mineola, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Shelby, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Rapid City, South Dakota
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Draper, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Salem, Virginia
- Czechia (3):
  - Research Site, Brno
  - Research Site, Pardubice
  - Research Site, Prague
- Research Site, Tallinn, Estonia
- Poland (2):
  - Research Site, Lodz
  - Research Site, Warsaw
- Puerto Rico (3):
  - Research Site, Carolina
  - Research Site, Cidra
  - Research Site, San Juan

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com